CLINICAL TRIAL: NCT00997074
Title: The Effect of Prophylactic Ibuprofen Versus Placebo on Pain Relief and Success Rates of Medical Abortion: A Double-blind Randomized Placebo Controlled Study
Brief Title: Efficacy Study of Prophylactic Ibuprofen Versus Placebo on Pain Relief and Success Rates of Medical Abortion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Daniel Seidman, Senior Physician, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHEBA-09-7253-DS-CTIL
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Pain; Pregnancy
Keywords: pain after abortion; abortion
MeSH Terms: conditions — Pain | interventions — Ibuprofen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ibuprofen (Experimental): the group will receive 2 tablets of ibuprofen 400 mg at the time of misoprostol administration. The information about the effect of the analgesics on the pain, and on the course of medical abortion, will be prospectively gathered from questionnaires completed by the study participants
  Interventions: Drug: ibuprofen
- placebo (No Intervention): this group will receive 2 placebo tablets together with the misoprostol

INTERVENTIONS:
Drug: ibuprofen — The most common side effect observed during medical abortion using mifepristone together with misoprostol is abdominal pain. The use of ibuprofen was not shown to interfere with the action of misoprostol to induce uterine contractions and pregnancy expulsion.
  Other Names: ibuprofen - Nonsteroidal anti-inflammatory drugs (NSAIDs)
  Arms: ibuprofen

SUMMARY:
In the current study, we want to evaluate the prophylactic use of ibuprofen versus a placebo for medical abortion by mifepristone and misoprostol, at a gestational age of up to 7 weeks, in regard to the effect on pain relief and the overall procedure success.

expected results:

The prophylactic use of NSAIDs could offer significant pain relief and thereby a reduction in the need for additional pain relievers compared to the placebo, without interfering with the outcome of medical abortion

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Pregnancy of up to 7 weeks gestation.
* Approval from the Ministry of Health committee for termination of pregnancy after an intrauterine pregnancy was demonstrated by an ultrasound exam.
* Subjects that provided informed consent and agree to comply with all study procedures.

Exclusion Criteria:

* Known allergy to mifepristone, misoprostol, paracetamol or NSAIDs.
* Severe anemia.
* Drug or alcohol abuse
* Known abnormal liver function (liver function tests greater than 1.5 times upper range of normal).
* Known abnormal renal function (serum creatinine > 1.5 mg/dl).
* Abnormal blood tests
* Exclusionary health problems contraindicating mifepristone included adrenal disease; sickle cell anemia; severe liver, respiratory, or renal disease; and blood clotting defect.
* Chronic disease
* Patient is participating currently in another clinical trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
• Decrease in pain as assessed using an 11-point numeric pain scale from 0 (= no pain) to 10 (=most severe pain). | 2 weeks

SECONDARY OUTCOMES:
• Success of medical abortion as assessed by follow-up ultrasound examination and the frequency of surgical intervention was recorded. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Seidman, Prof., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Aviv, Israel

REFERENCES:
- [Result] Avraham S, Gat I, Duvdevani NR, Haas J, Frenkel Y, Seidman DS. Pre-emptive effect of ibuprofen versus placebo on pain relief and success rates of medical abortion: a double-blind, randomized, controlled study. Fertil Steril. 2012 Mar;97(3):612-5. doi: 10.1016/j.fertnstert.2011.12.041. Epub 2012 Jan 20. PMID 22265034
- [Derived] Reynolds-Wright JJ, Woldetsadik MA, Morroni C, Cameron S. Pain management for medical abortion before 14 weeks' gestation. Cochrane Database Syst Rev. 2022 May 13;5(5):CD013525. doi: 10.1002/14651858.CD013525.pub2. PMID 35553047